CLINICAL TRIAL: NCT05261035
Title: Effect of Stretching Exercises Versus Thermotherapy on Restless Legs Syndrome Symptoms, Pain, and Quality of Sleep Among Pregnant Women
Brief Title: Stretching Exercises Versus Thermotherapy on Restless Legs Syndrome Symptoms
Acronym: Exersize
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1206022021
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Muscle Disorder
Keywords: Muscle Stretching Exercises; Thermotherapy; Restless legs syndrome; Pain; Sleep quality; pregnant women
MeSH Terms: conditions — Muscular Diseases; Hyperthermia; Restless Legs Syndrome; Pain; Sleep Initiation and Maintenance Disorders | interventions — Muscle Stretching Exercises; Hyperthermia, Induced

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stretching exercises group (Experimental): Pregnant women with RLS were instructed to perform stretching exercises daily for one week
  Interventions: Behavioral: stretching exercises
- Thermotherapy group (Active Comparator): Pregnant women with RLS were instructed to apply warm water immersion of their legs daily for one week.
  Interventions: Other: thermotherapy

INTERVENTIONS:
Behavioral: stretching exercises — For the stretching exercises group; the researchers explained to the women how to perform the stretching exercises through different visual materials like videos & pictures, provided a demonstration of each step, and emphasized that they could perform this exercise at any comfortable position, standing, sitting, or dorsal.
  Arms: stretching exercises group
Other: thermotherapy — women were instructed to warm the water to 43-47 C° using a water thermometer or test it with the inner aspect of their wrists. They are also advised to avoid using too hot or too cold water. Then immerse their legs for 20 minutes in the warm water at a h
  Arms: Thermotherapy group

SUMMARY:
To compare the effects of stretching exercises versus thermotherapy on RLS symptoms and sleep quality among pregnant women.

Research hypotheses:

* Pregnant women who perform leg stretching exercises exhibit lower RLS symptoms severity and pain level than those who applied thermotherapy.
* Pregnant women who perform leg stretching exercises exhibit higher sleep quality than those who applied thermotherapy.

DETAILED DESCRIPTION:
a quasi-experimental study was carried out at the antenatal outpatient clinic of XXXX. A sample of 60 pregnant women was randomly assigned to two groups. One group was instructed to perform stretching exercises daily for one week, and the other group applied thermotherapy. They rated their RLS symptoms, pain level, and sleep quality at baseline and after receiving interventions.

A convenience sampling of 60 pregnant women who fulfilled the following inclusion criteria was recruited: suffering from RLS according to the IRLSSG criteria during the third-trimester of a singleton pregnancy; rated restlessness severity greater than ten on the RLS Rating Scale, and compliant with an iron supplement. While, women who had a high-risk pregnancy, e.g., preeclampsia, diabetes, and placenta previa as well as had leg cramps, periodic limb movement disorder, leg edema, myalgia, peripheral neuropathy, leg injuries, and anxiety were excluded from the study.

Initially, the researchers approached the pregnant women of both groups in the waiting area of the antenatal clinic, established rapport, and collected the socio-demographic data and current pregnancy profile, Moreover, baseline RLS symptoms severity, pain, and women's sleep quality were assessed.

Interventions

For the stretching exercises group; the researchers explained to the women how to perform the stretching exercises through different visual materials like videos & pictures, provided a demonstration of each step, and emphasized that they could perform this exercise at any comfortable position, standing, sitting, or dorsal.

For the thermotherapy group, women were instructed to warm the water to 43-47 C° using a water thermometer or test it with the inner aspect of their wrists. They are also advised to avoid using too hot or too cold water. Then immerse their legs for 20 minutes in the warm water at a height where the water level can reach their knees. The researchers emphasized that the procedure should be done every night for one week.

For both groups, the intensity of RLS and pain severity of pregnant women of the two groups were reassessed after the first session.

ELIGIBILITY:
Inclusion Criteria:

* Had singleton pregnancy
* During the third-trimester
* Rated restlessness severity greater than ten on the RLS Rating Scale
* Compliant with an iron supplement.

Exclusion Criteria:

* Had a high-risk pregnancy
* Periodic limb movement disorder
* Leg edema
* Myalgia
* Peripheral neuropathy
* Leg injuries
* Anxiety

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
RLS Rating Scale | After 7 days
  This tool was adopted from the International RLS Study Group. The scale was designed to grade the severity of RLS symptoms. It is composed of ten items rated on a four-point Likert scale ranging from mild (1) to very severe (4). The total scores ranged from 10-to 40. The severity of women's restless leg symptoms was categorized as follows; very severe symptoms (scores 31- 40), Severe (scores 21- 30), Moderate (scores 11-20), Mild (scores 1-10). Abetz, et al. tested RLS Rating Scale for validity and reliability. The concurrent validity was r = 0.70, and internal consistency, alpha=0.81.16
Numeric Pain Rating Scale (NPRS) | After 7 days
  This tool was adopted from the Clinical Manual for Nursing Practice.17 It is a unidimensional measure of pain severity in adult individuals; the 11-point numeric scale varies from "0" (no pain) to "10" (severe pain). It was used to assess four levels of pain: 0 = no pain, 1-3= mild pain, 4-6 = moderate pain, 7-10 = severe pain.

SECONDARY OUTCOMES:
Groningen Sleep Quality Scale (GSQS) | After 7 days
  This scale is used to assess the subjects' sleeping patterns and overall sleep quality. It consists of 15-items that scored as true or false. One point was given for all the true items except items 8, 10, and 12 had reversed scores. The scoring system of this scale is as follows; the first question is not counted toward the total score therefore, scores ranged from 0 to 14. According to the total scores, the sleep quality was categorized into three categories; normal refreshing sleep "score 0-2", slightly disturbed sleep "scores 3-9", and poor quality of sleep "scores 10-14". In a validation study, the mean score on the scale was 6.0 ± 4.2 and Cronbach's alpha for internal consistency was 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen RP, Picchietti D, Hening WA, Trenkwalder C, Walters AS, Montplaisi J; Restless Legs Syndrome Diagnosis and Epidemiology workshop at the National Institutes of Health; International Restless Legs Syndrome Study Group. Restless legs syndrome: diagnostic criteria, special considerations, and epidemiology. A report from the restless legs syndrome diagnosis and epidemiology workshop at the National Institutes of Health. Sleep Med. 2003 Mar;4(2):101-19. doi: 10.1016/s1389-9457(03)00010-8. PMID 14592341
- [Background] Jafarimanesh H, Vakilian K, Mobasseri S. Thermo-therapy and cryotherapy to decrease the symptoms of restless leg syndrome during the pregnancy: A randomized clinical trial. Complement Ther Med. 2020 May;50:102409. doi: 10.1016/j.ctim.2020.102409. Epub 2020 Apr 19. PMID 32444058
- [Background] Sonmez A, Aksoy Derya Y. Effects of sleep hygiene training given to pregnant women with restless leg syndrome on their sleep quality. Sleep Breath. 2018 May;22(2):527-535. doi: 10.1007/s11325-018-1619-5. Epub 2018 Jan 13. PMID 29332218
- [Background] Darvishi N, Daneshkhah A, Khaledi-Paveh B, Vaisi-Raygani A, Mohammadi M, Salari N, Darvishi F, Abdi A, Jalali R. The prevalence of Restless Legs Syndrome/Willis-ekbom disease (RLS/WED) in the third trimester of pregnancy: a systematic review. BMC Neurol. 2020 Apr 13;20(1):132. doi: 10.1186/s12883-020-01709-0. PMID 32284042